CLINICAL TRIAL: NCT06781528
Title: Postpartum Hemorrhage and Alterations in Uterine Ecostructure
Status: Completed | Type: Observational
Sponsor: IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other)
Responsible Party: Sponsor
Other Study IDs: EPP1.0
Record Dates: First submitted 2024-12-03; First posted 2025-01-17 (Actual); Last update posted 2025-01-17 (Actual); Status verified 2024-10

CONDITIONS: Postpartum Hemorrhage
Keywords: endometrium-myometrium junctional zone
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hemorrhagic participants: Participants who deliver at the Division of Obstetrics and Prenatal Age Medicine at Sant'Orsola Polyclinic by vaginal delivery or cesarean section complicated by primary postpartum hemorrhage.
  Interventions: Other: Ultrasound evaluation
- No hemorrhagic participants: Participants who deliver at the Division of Obstetrics and Prenatal Age Medicine of Sant'Orsola Polyclinic by vaginal delivery or cesarean section not complicated by postpartum hemorrhage or other adverse obstetrical events matched for gestational age and parity at delivery.
  Interventions: Other: Ultrasound evaluation

INTERVENTIONS:
Other: Ultrasound evaluation — All patients will undergo 2D and 3D transvaginal ultrasonography 6-12 months after delivery at the outpatient clinics of our center, as per normal care procedure. Ultrasonographic evaluation aims to detect alterations of the uterine ecostructure, particularly of the endometrial-myometrial junctional zone. The presence of typical signs of uterine adenomyosis, in its various forms (diffuse, focal or localized-adenomyoma) will be investigated.

SUMMARY:
The goal of this observational study is to evaluate the presence of alterations in the ecostructure of the uterus in patients with a positive history of primary postpartum hemorrhage, in order to demonstrate a statistically significant correlation between these ecostructural alterations and adverse obstetric event.

DETAILED DESCRIPTION:
Over the past 10 years, numerous epidemiological studies have revealed an association between endometriosis and risk of adverse obstetrical events. Among the various mechanisms involved in the occurrence of some obstetrical diseases, alteration of endometrial/myometrial junction (JZ) would lead to abnormal trophoblastic invasion of the myometrial junctional zone due to partial or absent remodeling of uterine spiral arteries.

There are currently few studies in the literature on the topic, and those that do exist report conflicting results on the association between JZ alterations and risk of postpartum hemorrhage. Altered uterine contractile capacity and abnormal trophoblastic invasion of the myometrial endometrial junctional zone are the mechanisms called into question that could explain the increased risk of postpartum hemorrhage in patients. With this background, the purpose of our study is to highlight whether the presence of poor definition of the endometrial/myometrial junction, its thickening, or the presence in its context of irregularities and discontinuities represent a risk factor associated with the development of postpartum hemorrhage or are uterine ecostructural changes that develop consequent to a postpartum hemorrhage event.

All patients will be recruited during the puerperium stay at the Division of Obstetrics and Prenatal Age Medicine at Sant'Orsola Polyclinic. Subsequently, women will undergo gynecological examination and transvaginal ultrasound 6-12 months after delivery at the outpatient clinics of the same division.

In addition to the standard transvaginal gynecologic examination and ultrasonography, a 3D evaluation of the uterus and the endometrium-myometrium junctional zone will be performed using a Voluson E8 ultrasound machine (GE, Milan, Italy). This assessment will be quick and painless for the patient and it will last a maximum of five minutes.

For each patient, information will be collected on:

* Age
* Ethnicity
* Body mass index (BMI)
* Relevant pathologies
* Previous uterine surgery (myomectomy, CT scan, OCR)
* Associated symptoms: Dysmenorrhea, Chronic pelvic pain, Pain on ovulation, Dyspareunia, Dysuria, Dyschezia, Alterations in alvus, Abdominal bloating, Abnormal uterine bleeding (menometrorrhagia or spotting)
* Presence of uterine fibroids
* Presence of pelvic endometriosis
* Parity
* Mode of pregnancy onset (spontaneous vs. medically assisted procreation)
* Multiple pregnancy
* Any placental pathologies: placenta previa, accretism, suspected or established detachment.
* Any pathologies arising in pregnancy: gestational hypertension, preclampsia, diabetes
* Gestational age at the time of delivery
* Mode of delivery (vaginal/caesarean section)
* Neonatal weight
* Possible cervical, vulvo-vaginal tears.
* Abnormalities of secondment
* Uterine ultrasound features (classification according to MUSA study)

ELIGIBILITY:
Inclusion Criteria Group A:

* Age > 18 years
* Acquisition of Informed Consent Form
* Primary postpartum hemorrhage (defined as blood loss greater than or equal to 1 liter or blood loss that is accompanied by signs and symptoms of hypovolemia occurring within 24 hours of delivery)

Inclusion Criteria Group B:

* Age > 18 years
* Acquisition of Informed Consent Form
* Delivery not complicated by postpartum hemorrhage or other adverse obstetric events

Exclusion Criteria:

* Known uterine myomas or previous myomectomy surgery
* Presence of pelvic endometriosis
* Maternal hypertensive conditions
* Pluriparity (> 3)
* Multiple pregnancy
* Polydramnios
* Obesity (BMI> 35)
* Neonatal macrosomia
* Known coaugulopathies/thrombocytopenias
* Refusal to undergo subsequent follow-up at our center

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Group A will consist of patients who gave birth at the Division of Obstetrics and Prenatal Age Medicine at Sant'Orsola Polyclinic by vaginal delivery or cesarean section complicated by primary postpartum hemorrhage. Group B will consist of women who delivered at the same facility by vaginal delivery or cesarean section not complicated by postpartum hemorrhage or other adverse obstetric events matched for gestational age and parity at delivery.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-06-10 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Evaluation of the presence of changes in uterine ecostructure | 6-12 months after delivery
  Evaluation of the presence of alterations in the ecostructure of the uterus and in particular the endometrium-myometrium junctional zone (JZ) in patients with a positive history of primary postpartum hemorrhage, in order to demonstrate a statistically significant correlation between these ecostructural alterations and adverse obstetric event.

CONTACTS AND LOCATIONS:
Overall Officials: Gianluigi Pilu, MD, Principal Investigator — IRCCS Azienda Ospedaliero-Universitaria di Bologna
Locations (1):
- IRCCS Azienda Ospedaliero-Universitaria di Bologna, Bologna, Bologna, Italy